CLINICAL TRIAL: NCT03076996
Title: Youth Power Action Feasibility Study of Online Support Group Intervention Among Adolescents Living With HIV in Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 930307
Record Dates: First submitted 2017-02-08; First posted 2017-03-10 (Actual); Results first posted 2019-02-18 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: HIV/AIDS; Adolescent Behavior; Medication Adherence; Health Behavior
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Adolescent Behavior; Medication Adherence; Health Behavior

STUDY DESIGN:
Intervention Model Description: Single group pre/post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online support group (Experimental): Participants will be enrolled to receive six sessions from the Positive Connections curriculum through the m/eHealth intervention that will use Facebook to conduct online structured support groups.
  Interventions: Behavioral: Online support group

INTERVENTIONS:
Behavioral: Online support group — Participants will be enrolled to form five groups of 8 to 10 participants, and then participants will participate in the 6 sessions of the structured educational and group counseling curriculum through the online platform.
  The m/eHealth intervention components include:
  * Informational messages that reflect the content of the structured group counseling curriculum, Positive Connections, and are posted to the group wall on a regular basis
  * Moderated, closed group chats where ALHIV can interact with their peers and with a trained health counselor on a biweekly basis
  * Access to a trained counselor via Facebook Messenger (during normal business hours) for the duration of the intervention who will be able to provide information or basic counseling on ART/HIV care related issues, with referral to health care services as needed

SUMMARY:
This study will examine the feasibility and acceptability of an intervention designed to improve retention in HIV care services and improve anti-retroviral therapy (ART) adherence among adolescents ages 15-19 years living with HIV enrolled in ART services.

DETAILED DESCRIPTION:
Study aim is to examine the feasibility and acceptability of an intervention designed to improve retention in HIV care services and improve anti-retroviral therapy (ART) adherence among adolescents ages 15-19 years living with HIV enrolled in ART services.

A single group, pre/posttest design including structured questionnaires with adolescents living with HIV. Additionally, we will abstract clinical data from the medical record system. We will also conduct in-depth interviews with a subset of participants, as well as health care staff who are engaged in the intervention, at endline.

The objectives of this study are:

1. To examine the feasibility of implementing a mobile/electronic health (m/eHealth) intervention designed to improve retention in HIV care services and ART adherence among ALHIV ages 15-19 years through an online support group (using Facebook).
2. To assess acceptability of and engagement in the intervention by the target audience to inform improvements to the intervention.
3. To gather preliminary data on the psycho-social and health-related outcomes that the intervention is designed to affect to inform an outcome evaluation study that will be conducted following the conclusion of the feasibility study.
4. To collect information on recruitment, informed consent and data collection processes to inform the outcome evaluation study of the current intervention that will be conducted once findings from this feasibility study are incorporated into the intervention design.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive and currently on ART for at least 6 months
* Age 15 to 19 years
* Can demonstrate basic literacy necessary to participate in online chats

Exclusion Criteria:

* Not planning to remain in the study area (within Akwa Ibom State) for the duration of the study (approximately 6 months)
* Currently enrolled in an in-person support group
* Currently enrolled in another research study related to HIV service retention or ART adherence
* Critically or severely ill requiring hospitalization or such that the individual is unable to provide informed consent at the time of study recruitment

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Dulli, PhD, Principal Investigator — FHI 360
Locations (1):
- SIDHAS-supported facilities, Uyo, Always Ibom, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dulli L, Ridgeway K, Packer C, Plourde KF, Mumuni T, Idaboh T, Olumide A, Ojengbede O, McCarraher DR. An Online Support Group Intervention for Adolescents Living with HIV in Nigeria: A Pre-Post Test Study. JMIR Public Health Surveill. 2018 Nov 28;4(4):e12397. doi: 10.2196/12397. PMID 30487116

RESULTS

PARTICIPANT FLOW:
Groups:
- Online Support Group: Intervention content was delivered online through "secret" Facebook groups that limit membership and access to those invited and added by a group administrator. Intervention components included informational messages and moderated group discussions. Five sessions were included: 1) Understanding HIV; 2) Disclosure and Developing Trust in Relationships; 3) Treatment and Adherence; 4) Nutrition and Health; and 5) Sex and Relationships. Sessions activities included: 1) At-a-glance, introducing the topic of the week; 2) Word of the week, defining one key concept for the topic; 3) Cartoons used to tell a story related to the topic; 4) Key messages to deliver important information; 5) Quizzes to assess participants' knowledge and stimulate discussion; and 6) Group discussions moderated by facilitators. Groups began with an initial, in-person meeting. All participants received a basic cellular phone that could access Facebook, regardless of current phone ownership.
Period: Overall Study
Arm/Group | Online Support Group
Started | 41
Completed | 35
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 3
Not completed — Literacy precluded participation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Online Support Group
Number analyzed (Participants) | 41
Age, Continuous [Mean (Full Range); unit: Years] | 17 [15 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Nigeria | 41
religion [Count of Participants; unit: Participants]
  Catholic | 1
  All other Christian | 40
Time on ART [Mean (Full Range); unit: Years] | 3.8 [0.5 to 10.9]
Education [Count of Participants; unit: Participants]
  Currently enrolled in school, junior or secondary | 5
  Currently enrolled in school, post-secondary | 15
  Not currently enrolled, completed some secondary | 6
  Not currently enrolled, complete secondary | 15
Currently employed [Count of Participants; unit: Participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Active Members Who Have at Least One Post in Group Chat Session.
Description: Participants level of engagement in support group activities informs on the feasibility of intervention, measured by percentage of active members who have at least one post in group chat session.
Time Frame: 3 months
Population: Participants who initiated the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Online Support Group
Number analyzed (Participants) | 38
Participants | 32

2. Secondary Outcome: Acceptability Score
Description: Acceptability score: A set of ten items asking if participants agreed=1 or disagreed=0 with statements on acceptability. Score represents a sum of the 10 items with a range of 0 to 10, and a greater number indicating agreement with more acceptability items.
Time Frame: 3 months
Population: Endline participants who participated in the intervention
Measure: Mean (Full Range); unit: Scores on Scale
Arm/Group | Online Support Group
Number analyzed (Participants) | 34
Scores on Scale | 9.9 [9 to 10]

3. Secondary Outcome: Adherence to ART as Measured by the AACTG Adherence Assessment
Description: Proportion of participants who report not having missed any ART doses in past 3 days.
Time Frame: 3 months
Population: Participants who completed end line questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Online Support Group
Number analyzed (Participants) | 35
Participants | 29

4. Secondary Outcome: Adherence to Follow-up Visit Within 1 Month of Scheduled Date
Description: Retention in HIV services will be measured using data abstracted from the medical record system on date of visits between enrollment and the endline of this study. To be considered retained in HIV services, an individual must, at 3 months after enrollment, have attended his/her most recently scheduled clinical follow-up visit within 1 month of the date when it was scheduled to take place.
Time Frame: 3 months
Population: Participants enrolled in study at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Online Support Group
Number analyzed (Participants) | 41
Participants | 37

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Online Support Group
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

LIMITATIONS AND CAVEATS:
The non-probability sample precludes generalizing results beyond the study sample.

Social desirability bias may play a role in participants' responses to questions about the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT03076996/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT03076996/SAP_001.pdf